CLINICAL TRIAL: NCT04433663
Title: Eating Disorders, Emotion Regulation, and Mentalization: Addressing the Gap Between Theory and Practice
Brief Title: Eating Disorders, Self Regulation and Mentalization
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tel Hai College (Other)
Responsible Party: Principal Investigator, Moria Golan, Prof., Tel Hai College
Allocation: Randomized | Model: Sequential | Masking: Triple | Purpose: Treatment
Other Study IDs: TelHaiC
Record Dates: First submitted 2020-05-31; First posted 2020-06-16 (Actual); Last update posted 2020-10-08 (Actual); Status verified 2020-10

CONDITIONS: Eating Disorders
Keywords: eating disorders; self-regulation; self-control; Mentalization
MeSH Terms: conditions — Feeding and Eating Disorders; Self-Control

STUDY DESIGN:
Intervention Model Description: Six experienced therapists (more than 10 yrs. in the eating disorders' treatment) within one eating disorder center, were randomly allocated using the excel randomization function to the intervention group and control group. All participants in the clinical sample were drawn consecutively from admitted population to these therapists in a community-based eating disorder center between September 2018 to April 2019.
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: The research student, who collected the data was blind to treatment groups. Therapists and participants were blinded to the research aims and hypothesis.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mentalization-based Intervention (Experimental): Participants in the intervention group, received mentalization-based psychotherapy with the developed ECOSA axis. Therapist received mentalization-based supervision.
  Interventions: Other: Mentalization -based therapy using novel tool to demonstrate eating behavior and control axis
- IPT-Inter Personal Therapy (Active Comparator): The control group's participants received IPT - interpersonal psychotherapy that focused on resolving interpersonal problems and symptomatic recovery. The control group's therapist received regular supervision - with no emphasis on mentalization or tool's usage.
  Interventions: Other: Mentalization -based therapy using novel tool to demonstrate eating behavior and control axis

INTERVENTIONS:
Other: Mentalization -based therapy using novel tool to demonstrate eating behavior and control axis — To address the gap between theory and practice in the treatment of eating disorders we y developed a novel axis, ECOSA, to better conceptualize the complex interaction between eating style, control conditions, and the impact of the "emotional brain" versus the "thinking brain". A randomized pilot study was used to evaluate the integration of this tool in a mentalization-based treatment compared to treatment as usual (IPT).
  Methods: The suggested tool was tested in a randomized blinded feasibility study using the Eating Attitudes Test (EAT-26) and the Reflective Functioning Questionnaire RFQ - as the main outcome.
  Other Names: IPT - interpersonal psychotherapy

SUMMARY:
A randomized blinded feasibility study using the Eating Attitudes Test (EAT-26) and the Reflective Functioning Questionnaire RFQ - as the main outcome to assess two interventions for eating disorders. Six experienced therapists, and their consecutively 8-9 admitted clients, were randomly allocated to the intervention group and control group. The sample included a total of 52 participants, all women, mean age 24.2 yrs. old. In the intervention group, participants received mentalization-based psychotherapy with ECOSA - a novel developed mentalization tool and in the control group, participants received interpersonal psychotherapy that focused on resolving interpersonal problems and symptomatic recovery. Four randomized samples for each participant were checked for therapy-focused fidelity by two different psychotherapists.

DETAILED DESCRIPTION:
Six experienced therapists (more than 10 yrs. in the eating disorders' treatment) within one eating disorder center, were randomly allocated using the excel randomization function to the intervention group and control group. All participants in the clinical sample were drawn consecutively from admitted population to these therapists in a community-based eating disorder center between September 2018 to April 2019. The sample (total of 52 patients) included 26 participants in each group, all women, (mean age 24.2±3.2). Forty two percent of participants in each group were diagnosed with BN, 13% with BED, 35% with AN and 10% with ARFID. Thirty percent of participants in each group, also met criteria for borderline personality disorder on the SCID-II .The overall sample had predominantly high socioeconomic status.

Each therapist received a written consent from 8 to 9 clients to participate in the study and record all sessions. The research student, who collected the data was blind to treatment groups. Therapists and participants were blinded to the research aims and hypothesis.

In the intervention group, therapist received mentalization-based supervision along all participants' treatments, with the suggested tool and facilitated mentalization-focused therapy. The control group's participants received ITP-interpersonal psychotherapy that focused on resolving interpersonal problems and symptomatic recovery. The control group's therapist received regular supervision - with no emphasis on mentalization or tool's usage.

Participants' sessions were recorded over 12 months of treatment. Four randomized samples for each participant were checked for therapy-focused fidelity by two different psychotherapist Measures All participants underwent on entry a standard assessment of eating disorder, including a semi structured interview to measure co-morbid disorders, by experienced psychologist. Participants in both groups completed the Eating Attitudes Test (EAT-26) and the Reflective Functioning Questionnaire RFQ as part of a larger assessment battery.

The EAT-26 is a self-administered questionnaire that reveals abnormal eating behaviors. It consists of 26 items with six components scored from 0 to 3 (Zero: "Never," "Rarely," and "Sometimes"; 1: "Often"; 2: "Very often"; and 3: "Always"). The total score range from 0 to 78, and a score ≥ 20 is considered to represent abnormal eating attitudes or behaviors. The Cronbach's alpha in this study ranged between 0.75-0.90.

The RFQ was developed as a brief, easy-to-administer screening measure to assess severe impairments or imbalances in mentalization capacities. It includes 8 items scaled on 7-point Likert-type scale scored from 0 to 3. High values on this scale indicate high uncertainty about mental states, hence difficulties with mentalizing. The Cronbach's alpha in this study ranged between 0.8-0.94.

Statistical analysis All analyses were conducted using SPSS 23®. Normality distributions and outliers for each outcome variable were examined prior to commencing analysis. Independent T-tests analysis was used to assess differences between groups at baseline and between groups' improvements. Paired T-tests within each group used to assess the improvement between baseline, and 12 months treatment. Pearson correlations were computed to assess the relationship between change in eating disorder's symptoms and change in mentalizing capacities.

ELIGIBILITY:
Inclusion criteria:

* Participants were previously diagnosed with eating disorder (Eat-26>21)
* 17 yrs age and older
* no acute suicidality
* no physical risks due to eating disorder's symptoms

Exclusion criteria:

* age <17 yrs old
* refusal to corporate with treatment
* Need of 24 hrs medical care

Ages: 17 Years to 30 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 52 (Actual)
Dates: Start 2018-09-02 (Actual); Primary Completion 2019-04-30 (Actual); Study Completion 2020-05-01 (Actual)

PRIMARY OUTCOMES:
Reflective Functioning Questionnaire RFQ | 1 year
  The RFQ was developed as a brief, easy-to-administer screening measure to assess severe impairments or imbalances in mentalization capacities. It includes 8 items scaled on 7-point Likert-type scale scored from 0 to 3. High values on this scale indicate high uncertainty about mental states, hence difficulties with mentalizing (Fonagy, Luyten, Moulton-Perkins, Lee, Warren et al, 2016). The Cronbach's alpha in this study ranged between 0.8-0.94.
Eating Attitudes Test (EAT-26) | 1 year
  The EAT-26 is a self-administered questionnaire that reveals abnormal eating behaviors. It consists of 26 items with six components scored from 0 to 3 (Zero: "Never," "Rarely," and "Sometimes"; 1: "Often"; 2: "Very often"; and 3: "Always"). The total score range from 0 to 78, and a score ≥ 20 is considered to represent abnormal eating attitudes or behaviors (Garner, 1991). The Cronbach's alpha in this study ranged between 0.75-0.90.

CONTACTS AND LOCATIONS:
Locations (1):
- Academic College of Tel Hai, Kiryat Shmona, North of Israel, Israel

IPD SHARING:
Plan to Share IPD: No
All names and identification data will be omitted from the file that will be sent to statistical assessments.

REFERENCES:
- [Background] Fonagy, P., Gergely, G., Jurist, E. L., & Target, M. (2018). Affect regulation, mentalization and the development of the self. Taylor and Francis Inc. https://doi.org/10.4324/9780429471643
- [Background] Fonagy P, Luyten P, Moulton-Perkins A, Lee YW, Warren F, Howard S, Ghinai R, Fearon P, Lowyck B. Development and Validation of a Self-Report Measure of Mentalizing: The Reflective Functioning Questionnaire. PLoS One. 2016 Jul 8;11(7):e0158678. doi: 10.1371/journal.pone.0158678. eCollection 2016. PMID 27392018
- [Background] Garner, D. (1991). The Eating Disorder Inventory-2: Professional Manual. Odessa, Florida: Psychological Assessment Resources.
- [Background] Juarascio, A., Manasse, S., Clark, K. E., Schaumberg, K., Kerrigan, S., Goldstein, S. P., & Forman, E. (2020). Understanding the overlap and differences in terms describing patterns of maladaptive avoidance and intolerance of negative emotional states. Personality and Individual Differences. Elsevier Ltd. https://doi.org/10.1016/j.paid.2020. 109859.